CLINICAL TRIAL: NCT01379326
Title: The Efficacy of a Single-dose Mebendazole Against Soil-transmitted Helminths in School Children
Brief Title: Monitoring the Efficacy of Anthelmintics for the Treatment of Soil Transmitted Helminths P2
Acronym: ConWorm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Commonwealth Scientific and Industrial Research Organisation, Australia (Other Government); World Health Organization (Other); Institut Pasteur, Cambodia (Other); The University of Queensland (Other); Oswaldo Cruz Foundation (Other); University of Nottingham (Other); University of Yaounde 1 (Other); Ivo de Carneri, Pemba Island, Tanzania (Unknown); National Institute of Malariology, Parasitology and Entomology, Vietnam (Other Government); Jimma University (Other); Fundación Huésped (Other); Queensland Institute of Medical Research (Other); Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/374
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Ascaris Lumbricoides; Ascaris Suum; Trichuris Trichiura; Trichuris Vulpis; Ancylostoma Duodenal; Ancylostoma Caninum; Ancylostoma Ceylanicum; Necator Americanus
MeSH Terms: conditions — Trichuriasis | interventions — Mebendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mebendazole (Experimental)
  Interventions: Drug: Mebendazole

INTERVENTIONS:
Drug: Mebendazole — All children providing stool samples will be treated with mebendazole single table of 500mg under supervision (chewing + water).

SUMMARY:
Objectives:

The overall objective is to monitor efficacy of mebendazole (MBZ) against Soil-Transmitted Helminths (STH).

The primary objective is:

(1) to monitor the efficacy a single dose 500 mg of mebendazole (MBZ) against Soil-Transmitted Helminths (STH) infections by means of Faecal Egg Count Reduction (FECR) and Cure Rate (CR).

The secondary objectives are:

1. to assess the occurrence of Necator americanus and Ancylostoma duodenal.
2. to assess the occurrence of β-tubulin mutations related to resistance before and after drug administration.
3. to evaluate the role of dogs and pigs as reservoir for zoonotic transmission.

DETAILED DESCRIPTION:
Primary objective:

Following obtaining informed consent, schoolchildren in the target age range group will be recruited and asked to provide a recent stool sample (an interval of less than 4 hours) that will be processed to determine the Faecal Egg Count (FEC) for each Soil-Transmitted Helminths (STH) present. For the initial sampling the aim is to enroll at least 250 infected children for at least one of the Soil-Transmitted Helminths (STH). This sample size was selected based on statistical analysis of study power, using random simulations of correlated over-dispersed Faecal Egg Count data reflecting the variance-covariance structure in a selection of real Faecal Egg Count (FEC) data sets. This analysis suggested that a sample size of up to 200 individuals (α = 0.05, power = 80%) was required to detect a 10 percentage point drop from a null efficacy of ~ 80% (mean percentage FEC ∆ per individual) over a wide range of infection scenarios. Standard power analyses for proportions also indicated that the detection of a ~10 percentage point drop from a null cure rate required sample sizes up to 200 (the largest samples being required to detect departures from null efficacies of around 50%). Given an anticipated non-compliance rate of 25%, a sample of 250 infected subjects was therefore considered necessary at each study site.

All children providing stool samples will be treated with mebendazole (MBZ) single table of 500mg under supervision (chewing + water). The mebendazole (MBZ) will be provided (free) by the coordinating group. Seven up to fourteen days (maximum interval) after treatment a second faecal sample will be collected from the children to determine again FEC. Subjects who are unable to provide a stool sample at follow-up, or who are experiencing a severe concurrent medical condition or have diarrhea at time of the first sampling, will be excluded from the study.

Secondary objectives:

In 5 study sites, faecal samples of 100 infected subjects should be preserved before treatment with mebendazole (MBZ) in one tube (1 gram in 10 ml 70% ethanol). Samples of the same children should be also preserved again in one tube (1 gram in 10 ml 70% ethanol) after treatment. Samples have be send to the Laboratory of Parasitology, Ghent University.

The samples, collected before and after treatment will be subsequently examined by molecular assays the occurrence Necator americanus/Ancylostoma duodenal and the occurrence of β-tubulin mutations related to resistance.

The samples collected before treatment will be subsequently examined by molecular assays to assess the role of animals as a reservoir for human Soil-Transmitted Helminths (STH).

Parasitological techniques, determination of Faecal Egg Count of Soil-Transmitted Helminths (STH). All fecal samples were processed using the McMaster egg counting technique for the detection and the enumeration of infections with A. lumbricoides, T. trichiura and hookworms. All study sites are familiar with the technique and McMaster slides were provided previously.

Molecular assays (Laboratory of Parasitology, Ghent University)and Deoxyribonucleic acid (DNA) extraction.

DNA of Soil-Transmitted Helminths (STH) will be extracted from the samples preserved in ethanol 70% using the Qiagen mini stool kit.

Molecular identification of Soil-Transmitted Helminths (STH). The presence of the Soil-Transmitted Helminths species: Ascaris (n= 2), Trichuris (n = 2) and hookworms (n = 4) will be assessed using different molecular assays. For the differentiation of Trichuris species, species-specific polymerase chain reaction (PCR) will be applied. For the differentiation of Ascaris and the canine hookworms a PCR-Restriction Fragment Length Polymorphism (PCR-RFLP) will be used. For the human hookworms, a quantitative PCR will be applied.

Presence of mutations in β-tubulin related to mebendazole (MBZ) resistance This specific objective will be performed in collaboration with McGill University (Canada).

Statistical analysis. Both Cure Rate (CR) and Faecal Egg Count Reduction (FECR) will be considered to monitor to efficacy of mebendazole (MBZ) against Soil-Transmitted Helminths. The statistical analysis will be assessed as described by Vercruysse et al., 2011.

ELIGIBILITY:
Exclusion Criteria:

* Subjects who are unable to provide a stool sample at follow-up
* Subjects who are experiencing a severe concurrent medical condition
* Subjects with diarrhea at first sampling

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Reduction of fecal egg counts at 14 days post-intervention. | At 14 days post-intervention.
  Fecal egg counts at intervention and at 14 days follow-up.

SECONDARY OUTCOMES:
Distribution of hookworms species. | Samples will be collected at 14 days of follow-up.
  Presence of zoonotic Soil-Transmitted Helminths species, mutations linked with anthelminthic resistance.

CONTACTS AND LOCATIONS:
Locations (9):
- Fundacion Huesped, Buenos Aires, Argentina
- Australia (2):
  - Commonwealth Scientific and Industrial Research Organisation, Brisbane
  - Queensland Institute for Medical Research, University of Queensland, Herston QLD
- Fundação Oswaldo Cruz, Belo Horizonte, Brazil
- Institut Pasteur in Cambodia, Clinical Pathology Unit, Phnom Penh, Cambodia
- University of Yaoundé I, Yaoundé I, Cameroon
- College of Public Health and Medical Sciences, Jimma University, Jimma, Ethiopia
- Ivo de Carneri, Pemba Island, Zanzibar, Tanzania
- National Institute for Malariology, Parasitology and Entomology, Hanoi, Vietnam

REFERENCES:
- [Derived] Levecke B, Montresor A, Albonico M, Ame SM, Behnke JM, Bethony JM, Noumedem CD, Engels D, Guillard B, Kotze AC, Krolewiecki AJ, McCarthy JS, Mekonnen Z, Periago MV, Sopheak H, Tchuem-Tchuente LA, Duong TT, Huong NT, Zeynudin A, Vercruysse J. Assessment of anthelmintic efficacy of mebendazole in school children in six countries where soil-transmitted helminths are endemic. PLoS Negl Trop Dis. 2014 Oct 9;8(10):e3204. doi: 10.1371/journal.pntd.0003204. eCollection 2014 Oct. PMID 25299391